CLINICAL TRIAL: NCT01636583
Title: Zinc Absorption From Enriched Drinking Water Compared With the Zinc Absorption From a Fortified Maize Pudding in Healthy Young Adults.
Brief Title: Zinc Absorption From Fortified Water
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Principal Investigator, Prof. Michael B. Zimmermann, Prof. Dr.med., Swiss Federal Institute of Technology
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HNL/CTC_LSFZn
Record Dates: First submitted 2012-06-29; First posted 2012-07-10 (Estimated); Last update posted 2012-11-08 (Estimated); Status verified 2012-11

CONDITIONS: Fractional Absorption of Zinc (Focus of the Study)
Keywords: zinc; absorption; bio-availability; aqueous zinc; zinc deficiency; zinc fortification
MeSH Terms: interventions — Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- LSF water without meal (Experimental): Composition of test meal: 67Zn-labelled LSF-fortified water (1 mg 67Zn as ZnSO4 + 1 mg of eluted Zn from LSF device of natural isotopic composition)
  Interventions: Device: LSF water without meal
- LSF water and inhibitory meal (Active Comparator): Composition of test meal: Maize porridge and 67Zn-labelled LSF-fortified water (1 mg 67Zn as ZnSO4 + 0.44 mg of eluted Zn from LSF device of natural isotopic composition)
  Interventions: Device: LSF water and inhibitory meal
- Fortified inhibitory meal with water (Active Comparator): Composition of test meal: Maize porridge (1 mg 67Zn as ZnSO4 + 0.44 mg Zn as ZnSO4 of natural isotopic composition) and high purity water
  Interventions: Other: Fortified inhibitory meal with water

INTERVENTIONS:
Device: LSF water without meal — Composition of test meal: 67Zn-labelled LSF-fortified water (1 mg 67Zn as ZnSO4 + 1 mg of eluted Zn from LSF device of natural isotopic composition)
  Arms: LSF water without meal
Device: LSF water and inhibitory meal — Composition of test meal: Maize porridge and 67Zn-labelled LSF-fortified water (1 mg 67Zn as ZnSO4 + 0.44 mg of eluted Zn from LSF device of natural isotopic composition)
  Arms: LSF water and inhibitory meal
Other: Fortified inhibitory meal with water — Composition of test meal: Maize porridge (1 mg 67Zn as ZnSO4 + 0.44 mg Zn as ZnSO4 of natural isotopic composition) and high purity water
  Arms: Fortified inhibitory meal with water

SUMMARY:
A water purifying system, called LifeStrawFamily (LSF), able to fortify water with zinc to a concentration of 4 mg/l has been developed. The aim of this study is to investigate whether the LSF strategy is advantageous in terms of zinc absorption compared to food fortification. This study wants to demonstrate whether aqueous zinc produced by the LSF device consumed within or outside meals is better absorbed than zinc from an enriched cereal-based staple food in healthy adults. In addition, the zinc absorption from the LSF-enriched water and from a fortified inhibitory cereal-based pudding will be compared.

DETAILED DESCRIPTION:
Zinc bioavailability from a food or diet depends on the content of zinc and the presence of inhibitors of zinc absorption, e.g. inositol phosphate, also known as phytic acid (PA), and it is typically estimated with the phytate to zinc molar ratio (Phy:Zn). A zinc absorption of 10-15% is estimated from diets containing mainly unrefined cereal grains or legumes with negligible amounts of animal proteins, which are dominant in developing countries (characterised by a Phy:Zn > 15). For comparison, a mixed animal and plant product diet (Phy:Zn ranging 5-15) is estimated to have an average zinc bioavailability of 20-30% whereas a diet with ample refined cereals and rich in animal foods (Phy:Zn < 5) would have average zinc bioavailability of 30-50% (12, 19). Fractional absorption from aqueous zinc sulphate or zinc chloride solutions taken in a fasting state has been shown to range 56-74% for doses of 0.5-10 mg zinc (20-24) and decreasing to 37-62% for doses of 13-30.1 mg zinc (22, 24). Zinc from drinking water consumed away from meals appears to be substantially better absorbed than that from composite foods. Alternative strategies, designed for providing zinc through the water supply, could prove useful in the global effort to control zinc deficiency.

To investigate whether zinc eluted from Lifestraw Family® (LSF) device via its specific zinc delivery system is more bioavailable than zinc from fortified cereals as zinc sulphate, we will perform a human absorption study based on the double isotopic tracer ratio technique. The fractional absorption of zinc (FAZ) from LSF-fortified water consumed with or without food will be compared to the FAZ from a fortified cereal. This will allow quantifying zinc bioavailability from the LSF eluted zinc 1) when LSF-water is consumed in fasting state 2) when LSF-water is consumed together with other foods 3) to compare the latter two with zinc absorption from a zinc fortified cereal.

The results of this study will provide information on the potential advantages of LSF fortification over zinc food fortification, which is currently the recommended delivery vehicle for zinc in country fortification programs (25, 26). Furthermore, comparing zinc bioavailability from LSF-water consumed alone or in combination with food will instruct about the optimal way to consume it. This information can be used to optimally design the delivery strategy in the planned efficacy trials. In the future, this information could also be integrated in the information recommendations for use for prospective end-consumers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of 18 to 45 years old
* Body Mass Index in the range of 19 to 25
* No mineral and vitamin supplements two weeks prior to the study and during the whole duration of the study
* Signed informed consent

Exclusion Criteria:

* Any metabolic, gastrointestinal or chronic disease (according to the subjects own statement)
* Long-term medication during the whole study (except for contraceptives
* Vegans
* Smoking
* Pregnancy
* Lactating
* Intention to become pregnant during the course of the study
* Lack of safe contraception, defined as:
* Female subjects of childbearing potential, not using and not willing to use a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator in individual cases.
* Consumption of mineral and vitamin supplements within 2 weeks prior to 1st test meal administration
* Earlier participation in any nutrition study using Zn stable isotopes as well as participation in any other clinical study within the last 30 days and during this study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2012-06; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Fractional absorption (FA) of oral zinc isotope | At baseline (day 1) and day 5.
  A spot urine sample will be collected at baseline (day 1) and 96+/-3 hours (at day 5) after test meal administration and will be used to quantify zinc FA from the test meal. The FA from the zinc enriched LSF water consumed with and without food will be compared with the FA from the zinc fortified cereal.

SECONDARY OUTCOMES:
Plasma zinc (PZn) | day 1
  Plasma zinc (PZn)concentration in blood samples will be analysed. PZn will be used to indicate if a participant is zinc deficient and therefore its absorption value from the test meals have to be treated with caution. PZn values will be compared to the corresponding cut-off values.
C-reactive protein (CRP) | day 1
  C-reactive protein (CRP) concentration in blood samples will be analysed. CRP will indicate the inflammation/infection status of the subject at time of screening. Inflammation/infection is a confounder of zinc deficiency.

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Zimmermann, MD, Study Chair — ETH, Laboratory of Human Nutrition; Diego Moretti, Dr., Principal Investigator — ETH, Laboratory of Human Nutrition
Locations (1):
- Clinical Trials Center, University Hospital, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Galetti V, Kujinga P, Mitchikpe CE, Zeder C, Tay F, Tossou F, Hounhouigan JD, Zimmermann MB, Moretti D. Efficacy of highly bioavailable zinc from fortified water: a randomized controlled trial in rural Beninese children. Am J Clin Nutr. 2015 Nov;102(5):1238-48. doi: 10.3945/ajcn.115.117028. Epub 2015 Oct 14. PMID 26468121